CLINICAL TRIAL: NCT04515147
Title: COVID-19: A Phase 2a, Partially Observer-blind, Multicenter, Controlled, Dose-confirmation Clinical Trial to Evaluate the Safety, Reactogenicity and Immunogenicity of the Investigational SARS-CoV-2 mRNA Vaccine CVnCoV in Adults >60 Years of Age and 18 to 60 Years of Age
Brief Title: A Dose-Confirmation Study to Evaluate the Safety, Reactogenicity and Immunogenicity of Vaccine CVnCoV in Healthy Adults for COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CureVac (Industry)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: CV-NCOV-002
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Coronavirus; Covid19; SARS-CoV-2; Severe Acute Respiratory Syndrome
Keywords: Vaccine; SARS; COVID; Safety; Reactogenicity; Immunogenicity
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Severe Acute Respiratory Syndrome | interventions — CVnCoV COVID-19 vaccine; Hepatitis A Vaccines; Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Part 1, Group 1: CVnCoV 6 μg (Experimental): Participants will be vaccinated with CVnCoV on Day 1 and Day 29. Participants in this group will be aged between 18 and 60 years old.
  Interventions: Biological: CVnCoV 6 μg
- Part 1, Group 2: CVnCoV 6 μg (Experimental): Participants will be vaccinated with CVnCoV on Day 1 and Day 29. Participants in this group will be aged over 60 years old.
  Interventions: Biological: CVnCoV 6 μg
- Part 1, Group 3: CVnCoV 12 μg (Experimental): Participants will be vaccinated with CVnCoV on Day 1 and Day 29. Participants in this group will be between the ages of 18 to 60 years old.
  CVnCoV will be administered again as a booster vaccination on Day 180 in a sub-group of participants.
  Interventions: Biological: CVnCoV 12 μg
- Part 1, Group 4: CVnCoV 12 μg (Experimental): Participants will be vaccinated with CVnCoV on Day 1 and Day 29. Participants in this group will be aged over 60 years old.
  CVnCoV will be administered again as a booster vaccination on Day 57 or Day 180 in a sub-group of participants.
  Interventions: Biological: CVnCoV 12 μg
- Part 1, Group 5: Hepatitis A vaccine (Active Comparator): Participants will be vaccinated with a hepatitis A vaccine on Day 1 and Day 29. Participants in this group will be aged between 18 and 60 years old.
  Interventions: Biological: Hepatitis A vaccine
- Part 1, Group 6: Pneumococcal vaccine (Active Comparator): Participants will be vaccinated with a pneumococcal vaccine on Day 1 and Day 29. Participants in this group will be aged over 60 years old.
  Interventions: Biological: Pneumococcal vaccine
- Part 2, Group 1: CVnCoV 12 µg (Experimental): Participants will be vaccinated with CVnCoV 12 µg on Day 1 and Day 29. Participants in this group will be aged between 18 and 60 years old.
  Interventions: Biological: CVnCoV 12μg
- Part 2, Group 2: Hepatitis A vaccine (Active Comparator): Participants will be vaccinated with a hepatitis A vaccine on Day 1 and Day 29. Participants in this group will be aged between 18 and 60 years old.
  Interventions: Biological: Hepatitis A vaccine
- Part 2, Group 3: CVnCoV 12 µg (Experimental): Participants will be vaccinated with CVnCoV 12 µg on Day 1 and Day 29. Participants in this group will be aged over 60 years old.
  Interventions: Biological: CVnCoV 12μg
- Part 2, Group 4: Pneumococcal vaccine (Active Comparator): Participants will be vaccinated with a pneumococcal vaccine on Day 1 and Day 29. Participants in this group will be aged over 60 years old.
  Interventions: Biological: Pneumococcal vaccine

INTERVENTIONS:
Biological: CVnCoV 6 μg — Participants will receive an intramuscular injection by needle in the deltoid area.
  Other Names: CV07050101
  Arms: Part 1, Group 1: CVnCoV 6 μg; Part 1, Group 2: CVnCoV 6 μg
Biological: CVnCoV 12 μg — Participants will receive an intramuscular injection by needle in the deltoid area.
  Other Names: CV07050101
  Arms: Part 1, Group 3: CVnCoV 12 μg; Part 1, Group 4: CVnCoV 12 μg
Biological: Hepatitis A vaccine — Participants will receive an intramuscular injection by needle in the deltoid area.
  Arms: Part 1, Group 5: Hepatitis A vaccine; Part 2, Group 2: Hepatitis A vaccine
Biological: Pneumococcal vaccine — Participants will receive an intramuscular injection by needle in the deltoid area.
  Arms: Part 1, Group 6: Pneumococcal vaccine; Part 2, Group 4: Pneumococcal vaccine
Biological: CVnCoV 12μg — Participants will receive an intramuscular injection by needle in the deltoid area.
  Other Names: CV07050101
  Arms: Part 2, Group 1: CVnCoV 12 µg; Part 2, Group 3: CVnCoV 12 µg

SUMMARY:
This study aims to evaluate the safety and reactogenicity profile after 1 and 2 dose administrations of investigational SARS-CoV-2 mRNA vaccine (CVnCoV) at different dose levels and to evaluate the humoral immune response after 1 and 2 dose administrations of CVnCoV.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants ≥18 years of age. A healthy participant is defined as an individual who is in good general health, according to the Investigator's assessment. Chronic health conditions are acceptable if the condition is considered well controlled with treatment according to the discretion of the Investigator.
* Expected to be compliant with protocol procedures and available for clinical follow-up through the last planned visit.
* Participants are able to understand and willing to provide informed consent.
* Physical examination without clinically significant findings according to the Investigator's assessment.
* Body mass index (BMI) ≥18.0 and ≤32.0 kg/m^2.
* Female participants of childbearing potential: at the time of enrollment, negative human chorionic gonadotropin (hCG) pregnancy test (serum) for female participants presumed to be of childbearing potential on the day of enrollment. On Day 1 (pre-vaccination): negative urine pregnancy test (required if serum pregnancy test was performed more than 3 days before).
* Female participants of childbearing potential must use highly effective methods of birth control from 2 weeks before the first administration of the trial vaccine until 3 months following the last administration. The following methods of birth control are considered highly effective when used consistently and correctly:

  * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal);
  * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable);
  * Intrauterine devices;
  * Intrauterine hormone-releasing systems;
  * Bilateral tubal occlusion;
  * Vasectomized partner;
  * Sexual abstinence (periodic abstinence [e.g., calendar, ovulation, symptothermal and post-ovulation methods] and withdrawal are not acceptable).
* Male participants should be instructed not to get their partners pregnant until 3 months after the last administration.

Exclusion Criteria:

* Use of any investigational or non-registered product (vaccine or drug) other than the trial vaccine within 28 days preceding the administration of the trial vaccine, or planned use during the trial period.
* Receipt of any other vaccines within 28 days prior to enrollment in this trial or planned receipt of any vaccine within 28 days of trial vaccine administration (primary dose or booster dose).
* Receipt of any investigational or licensed/authorized SARS-CoV-2 or other coronavirus vaccine prior to the administration of the trial vaccine.
* Any treatment with immunosuppressants or other immune-modifying drugs (including, but not limited to, corticosteroids, biologicals, and methotrexate) within 6 months prior to the administration of the trial vaccine or planned use during the trial, with the exception of topically-applied, inhaled, or intranasal steroids.
* Use of hormonal therapy for gender reassignment.
* Any medically diagnosed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination, including known human immunodeficiency virus infection, hepatitis B virus infection, and hepatitis C virus infection.
* History of immune-mediated or autoimmune disease.
* History of angioedema (known C1 inhibitor deficiency).
* History of anaphylaxis or allergy to any component of CVnCoV or aminoglycoside antibiotics.
* History of or current alcohol and/or drug abuse.
* Participants who are active smokers, were active smokers within the last year (including any vaping in the last year), or have a total smoking history ≥10 pack years. A pack year is calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked.
* History of virologically-confirmed Severe Acute Respiratory Syndrome (SARS), Middle East Respiratory Syndrome (MERS), or COVID-19 disease or known exposure (without any personal protective equipment) to an individual with confirmed COVID-19 disease or SARS-CoV-2 infection within the past 2 weeks.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of any dose of the trial vaccine.
* Presence or evidence of significant uncontrolled acute or chronic medical or psychiatric illness. Significant medical or psychiatric illnesses include but are not limited to:

  * Uncontrolled respiratory disease (e.g., chronic obstructive pulmonary disease, asthma), including use of the following asthma medications: intravenous corticosteroids, leukotriene modifiers, biologics.
  * Uncontrolled cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease, history of stroke, peripheral artery disease, pulmonary embolism).
  * History of myocarditis or pericarditis as an adult.
  * Diabetes mellitus (insulin-dependent).
  * Uncontrolled neurological disorders or Guillain-Barré syndrome or history of seizure, except for febrile seizures during childhood.
  * Current or past malignancy, unless completely resolved without sequelae for >5 years.
* Foreseeable non-compliance with protocol, as judged by the Investigator.
* For female participants: pregnancy or lactation.
* Participants with impaired coagulation or any bleeding disorder in whom an intramuscular injection or a blood draw is contraindicated. This includes participants on treatment with anticoagulants (e.g., vitamin K antagonists, novel oral anticoagulants, and heparin). Use of platelet aggregation inhibitors is not exclusionary.
* Participants employed by the Sponsor, Investigator, or trial site, or relatives of research staff working on this trial.
* Participants considered at the Investigator's discretion to be at increased risk of exposure to COVID-19 disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Centro de vacunación internacional - CEVAXIN Panama Clinic, Panama City, Panama
- Instituto de Investigación Nutricional, Lima, Peru

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was performed in Peru and Panama between 21 September 2020 and 21 February 2022.
Pre-assignment Details: Of the 1035 participants who were screened, 668 participants were enrolled and received trial vaccine.
Groups:
- CVnCoV 6 μg: Aged 18-60 Years: Participants in Part 1 were vaccinated with CVnCoV 6 μg as an intramuscular injection by needle in the deltoid area on Day 1 and Day 29. Participants in this group were aged between 18 and 60 years old.
- CVnCoV 6 μg: Aged >60 Years: Participants in Part 1 were vaccinated with CVnCoV 6 μg as an intramuscular injection by needle in the deltoid area on Day 1 and Day 29. Participants in this group were aged over 60 years old.
- CVnCoV 12 μg: Aged 18-60 Years: Participants in Part 1 and Part 2 were vaccinated with CVnCoV 12 μg as an intramuscular injection by needle in the deltoid area on Day 1 and Day 29. Participants in this group were between the ages of 18 to 60 years old.
  CVnCoV was administered again as a booster vaccination on Day 180 in a sub-group of participants in Part 1.
- CVnCoV 12 μg: Aged >60 Years: Participants in Part 1 and Part 2 were vaccinated with CVnCoV 12 μg as an intramuscular injection by needle in the deltoid area on Day 1 and Day 29. Participants in this group were aged over 60 years old.
  CVnCoV was administered again as a booster vaccination on Day 57 or Day 180 in a sub-group of participants in Part 1.
- Active Control - Hepatitis A Vaccine: Aged 18-60 Years: Participants in Part 1 and Part 2 were vaccinated with a hepatitis A vaccine as an intramuscular injection by needle in the deltoid area on Day 1 and Day 29. Participants in this group were aged between 18 and 60 years old.
- Active Control - Pneumococcal Vaccine: Aged >60 Years: Participants in Part 1 and Part 2 were vaccinated with a pneumococcal vaccine as an intramuscular injection by needle in the deltoid area on Day 1 and Day 29. Participants in this group were aged over 60 years old.
Period: Overall Study
Arm/Group | CVnCoV 6 μg: Aged 18-60 Years | CVnCoV 6 μg: Aged >60 Years | CVnCoV 12 μg: Aged 18-60 Years | CVnCoV 12 μg: Aged >60 Years | Active Control - Hepatitis A Vaccine: Aged 18-60 Years | Active Control - Pneumococcal Vaccine: Aged >60 Years
Started | 12 | 11 | 289 | 295 | 31 | 30
Completed | 11 | 10 | 274 | 268 | 28 | 20
Not Completed | 1 | 1 | 15 | 27 | 3 | 10
Not completed — Withdrawal by Subject | 1 | 0 | 10 | 18 | 1 | 8
Not completed — Lost to Follow-up | 0 | 1 | 5 | 6 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Miscellaneous | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All participants who received at least 1 dose of trial vaccine and for whom any post-vaccination safety data are available.
Groups:
- Total: Total of all reporting groups
Arm/Group | CVnCoV 6 μg: Aged 18-60 Years | CVnCoV 6 μg: Aged >60 Years | CVnCoV 12 μg: Aged 18-60 Years | CVnCoV 12 μg: Aged >60 Years | Active Control - Hepatitis A Vaccine: Aged 18-60 Years | Active Control - Pneumococcal Vaccine: Aged >60 Years | Total
Number analyzed (Participants) | 12 | 11 | 289 | 295 | 31 | 30 | 668
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (8.44) | 65.6 (4.08) | 38.1 (12.08) | 69.0 (6.06) | 31.6 (12.31) | 66.7 (5.07) | 53.4 (18.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 118 | 139 | 12 | 16 | 296
  Male | 5 | 7 | 171 | 156 | 19 | 14 | 372
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 11 | 283 | 287 | 31 | 30 | 654
  Not Hispanic or Latino | 0 | 0 | 6 | 8 | 0 | 0 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 0 | 0 | 3 | 10 | 0 | 1 | 14
  Black or African American | 0 | 0 | 2 | 1 | 1 | 0 | 4
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Other | 12 | 11 | 283 | 284 | 30 | 29 | 649

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Solicited Adverse Event (AE) Occurring on the Day of Vaccination and the Following 7 Days After Dose 1 and Dose 2
Description: Solicited local AEs (injection site pain, redness, swelling, and itching) and solicited systemic AEs (fever, headache, fatigue, chills, myalgia, arthralgia, nausea/vomiting, and diarrhea) were recorded on the day of vaccination and the following 7 days using a diary (electronic or paper). By definition, all solicited local AEs occurring from the time of first vaccination were considered related to trial vaccination. For solicited systemic AEs, the Investigator assessed the relationship between trial vaccine and each occurrence of each AE.
Time Frame: Up to 7 days after Dose 1 (Days 1 to 8) and Dose 2 (Days 29 to 36)
Population: Safety Analysis Set: All participants who received at least 1 dose of trial vaccine and for whom any post-vaccination safety data are available. Only participants with evaluable samples at each visit are included.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 6 μg: Aged 18-60 Years | CVnCoV 6 μg: Aged >60 Years | CVnCoV 12 μg: Aged 18-60 Years | CVnCoV 12 μg: Aged >60 Years | Active Control - Hepatitis A Vaccine: Aged 18-60 Years | Active Control - Pneumococcal Vaccine: Aged >60 Years
Number analyzed (Participants) | 12 | 11 | 289 | 295 | 31 | 30
Participants
  Dose 1: Any solicited local AEs | 9 | 5 | 253 | 220 | 17 | 26
  Dose 1: Any solicited systemic AEs | 4 | 6 | 229 | 193 | 13 | 14
  Dose 1: Any related solicited systemic AEs | 4 | 5 | 228 | 190 | 13 | 14
  Dose 2: Any solicited local AEs: number analyzed (Participants) | 12 | 11 | 264 | 281 | 28 | 28
  Dose 2: Any solicited local AEs | 9 | 3 | 208 | 188 | 6 | 22
  Dose 2: Any solicited systemic AEs: number analyzed (Participants) | 12 | 11 | 264 | 281 | 28 | 28
  Dose 2: Any solicited systemic AEs | 9 | 8 | 217 | 195 | 13 | 11
  Dose 2: Any related solicited systemic AEs: number analyzed (Participants) | 12 | 11 | 264 | 281 | 28 | 28
  Dose 2: Any related solicited systemic AEs | 8 | 8 | 217 | 193 | 13 | 11

2. Primary Outcome: Intensity of Solicited AEs Per US Food and Drug Administration (FDA) Toxicity Grading Scale Occurring on the Day of Vaccination and the Following 7 Days After Dose 1 and Dose 2
Description: Solicited local AEs (injection site pain, redness, swelling, and itching) and solicited systemic AEs (fever, headache, fatigue, chills, myalgia, arthralgia, nausea/vomiting, and diarrhea) were recorded on the day of vaccination and the following 7 days using a diary (electronic or paper). Intensity of solicited local AEs and solicited systemic AEs were graded per the FDA Toxicity Grading Scale at Grades 1-3, where higher grades indicate a worse outcome.
Time Frame: Up to 7 days after Dose 1 (Days 1 to 8) and Dose 2 (Days 29 to 36)
Population: The Safety Analysis Set including only participants who experienced solicited local and systemic AEs. Only participants with evaluable samples at each visit are included.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 6 μg: Aged 18-60 Years | CVnCoV 6 μg: Aged >60 Years | CVnCoV 12 μg: Aged 18-60 Years | CVnCoV 12 μg: Aged >60 Years | Active Control - Hepatitis A Vaccine: Aged 18-60 Years | Active Control - Pneumococcal Vaccine: Aged >60 Years
Number analyzed (Participants) | 9 | 8 | 253 | 220 | 17 | 26
Participants
  Dose 1: Any solicited local AEs: number analyzed (Participants) | 9 | 5 | 253 | 220 | 17 | 26
  Dose 1: Any solicited local AEs: Grade 1 | 9 | 5 | 191 | 203 | 16 | 25
  Dose 1: Any solicited local AEs: Grade 2 | 0 | 0 | 61 | 17 | 1 | 1
  Dose 1: Any solicited local AEs: Grade 3 | 0 | 0 | 1 | 0 | 0 | 0
  Dose 1: Any solicited systemic AEs: number analyzed (Participants) | 4 | 6 | 229 | 193 | 13 | 14
  Dose 1: Any solicited systemic AEs: Grade 1 | 4 | 4 | 122 | 122 | 7 | 11
  Dose 1: Any solicited systemic AEs: Grade 2 | 0 | 2 | 96 | 65 | 6 | 3
  Dose 1: Any solicited systemic AEs: Grade 3 | 0 | 0 | 11 | 6 | 0 | 0
  Dose 2: Any solicited local AEs: number analyzed (Participants) | 9 | 3 | 208 | 188 | 6 | 22
  Dose 2: Any solicited local AEs: Grade 1 | 9 | 2 | 166 | 162 | 5 | 17
  Dose 2: Any solicited local AEs: Grade 2 | 0 | 1 | 42 | 25 | 1 | 5
  Dose 2: Any solicited local AEs: Grade 3 | 0 | 0 | 0 | 1 | 0 | 0
  Dose 2: Any solicited systemic AEs: number analyzed (Participants) | 9 | 8 | 217 | 195 | 13 | 11
  Dose 2: Any solicited systemic AEs: Grade 1 | 7 | 5 | 100 | 103 | 7 | 8
  Dose 2: Any solicited systemic AEs: Grade 2 | 2 | 1 | 109 | 83 | 6 | 3
  Dose 2: Any solicited systemic AEs: Grade 3 | 0 | 2 | 8 | 9 | 0 | 0

3. Primary Outcome: Duration of Solicited AEs Occurring on the Day of Vaccination and the Following 7 Days After After Dose 1 and Dose 2
Description: Solicited local AEs (injection site pain, redness, swelling, and itching) and solicited systemic AEs (fever, headache, fatigue, chills, myalgia, arthralgia, nausea/vomiting, and diarrhea) were recorded on the day of vaccination and the following 7 days using a diary (electronic or paper). Duration is calculated as consecutive days with a respective solicited AE regardless of the grade of the AE. AEs ongoing after day 8 are included.
Time Frame: Up to 7 days after Dose 1 (Days 1 to 8) and Dose 2 (Days 29 to 36)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Groups:
- Active Control - Hepatitis A Vaccine: Aged 18-60 Years: Active Control - Participants in Part 1 and Part 2 were vaccinated with a hepatitis A vaccine as an intramuscular injection by needle in the deltoid area on Day 1 and Day 29. Participants in this group were aged between 18 and 60 years old.
- Active Control - Pneumococcal Vaccine: Aged >60 Years: Active Control - Participants in Part 1 and Part 2 were vaccinated with a pneumococcal vaccine as an intramuscular injection by needle in the deltoid area on Day 1 and Day 29. Participants in this group were aged over 60 years old.
Arm/Group | CVnCoV 6 μg: Aged 18-60 Years | CVnCoV 6 μg: Aged >60 Years | CVnCoV 12 μg: Aged 18-60 Years | CVnCoV 12 μg: Aged >60 Years | Active Control - Hepatitis A Vaccine: Aged 18-60 Years | Active Control - Pneumococcal Vaccine: Aged >60 Years
Number analyzed (Participants) | 9 | 8 | 253 | 220 | 17 | 26
days
  Dose 1: Any solicited local AEs: number analyzed (Participants) | 9 | 5 | 253 | 220 | 17 | 26
  Dose 1: Any solicited local AEs | 1.3 (0.50) | 1.2 (0.45) | 2.1 (1.12) | 1.8 (1.54) | 1.6 (0.87) | 2.0 (1.20)
  Dose 1: Any solicited systemic AEs: number analyzed (Participants) | 4 | 6 | 229 | 193 | 13 | 14
  Dose 1: Any solicited systemic AEs | 1.5 (1.00) | 1.5 (0.84) | 1.9 (1.25) | 2.1 (1.42) | 1.9 (0.86) | 2.4 (2.17)
  Dose 2: Any solicited local AEs: number analyzed (Participants) | 9 | 3 | 208 | 188 | 6 | 22
  Dose 2: Any solicited local AEs | 2.1 (1.27) | 2.3 (1.15) | 2.2 (1.11) | 1.9 (1.33) | 2.2 (1.17) | 2.2 (0.96)
  Dose 2: Any solicited systemic AEs: number analyzed (Participants) | 9 | 8 | 217 | 195 | 13 | 11
  Dose 2: Any solicited systemic AEs | 2.1 (2.32) | 2.3 (2.43) | 1.9 (1.13) | 2.1 (1.49) | 2.2 (2.45) | 2.3 (2.05)

4. Primary Outcome: Number of Participants Who Experienced an Unsolicited AE Occurring on the Day of Vaccination and the Following 28 Days After Dose 1 and Dose 2
Description: Diaries were used for collection of unsolicited AEs on each vaccination day and the following 28 days. In addition, participants received a prompt (by e.g., a phone call or text message) to verify whether the participants had any health concerns since the last visit. The Investigator assessed the relationship between trial vaccine and each occurrence of each AE.
Time Frame: Up to 28 days after Dose 1 (Days 1 to 29) and Dose 2 (Days 29 to 57)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 6 μg: Aged 18-60 Years | CVnCoV 6 μg: Aged >60 Years | CVnCoV 12 μg: Aged 18-60 Years | CVnCoV 12 μg: Aged >60 Years | Active Control - Hepatitis A Vaccine: Aged 18-60 Years | Active Control - Pneumococcal Vaccine: Aged >60 Years
Number analyzed (Participants) | 12 | 11 | 289 | 295 | 31 | 30
Participants
  Dose 1: Any unsolicited AEs | 5 | 6 | 120 | 105 | 7 | 5
  Dose 1: Any related unsolicited AEs | 2 | 1 | 33 | 26 | 0 | 1
  Dose 2: Any unsolicited AEs: number analyzed (Participants) | 12 | 11 | 264 | 281 | 28 | 28
  Dose 2: Any unsolicited AEs | 4 | 3 | 77 | 75 | 10 | 7
  Dose 2: Any related unsolicited AEs: number analyzed (Participants) | 12 | 11 | 264 | 281 | 28 | 28
  Dose 2: Any related unsolicited AEs | 1 | 2 | 13 | 7 | 1 | 2

5. Primary Outcome: Intensity of Unsolicited AEs Per the Investigator's Assessment Occurring on the Day of Vaccination and the Following 28 Days After Dose 1 and Dose 2
Description: Diaries were used for collection of unsolicited AEs on each vaccination day and the following 28 days. In addition, participants received a prompt (by e.g., a phone call or text message) to verify whether the participants had any health concerns since the last visit. The Investigator made an assessment of intensity for each AE reported during the trial and assigned it to one of the following categories:
  * Mild: an event that was easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities.
  * Moderate: an event that caused sufficient discomfort to interfere with normal everyday activities.
  * Severe: an event that prevented normal everyday activities.
Time Frame: Up to 28 days after Dose 1 (Days 1 to 29) and Dose 2 (Days 29 to 57)
Population: The Safety Analysis Set including only participants who experienced unsolicited AEs. Only participants with evaluable samples at each visit are included.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 6 μg: Aged 18-60 Years | CVnCoV 6 μg: Aged >60 Years | CVnCoV 12 μg: Aged 18-60 Years | CVnCoV 12 μg: Aged >60 Years | Active Control - Hepatitis A Vaccine: Aged 18-60 Years | Active Control - Pneumococcal Vaccine: Aged >60 Years
Number analyzed (Participants) | 5 | 6 | 120 | 105 | 10 | 7
Participants
  Dose 1: Unsolicited AEs: number analyzed (Participants) | 5 | 6 | 120 | 105 | 7 | 5
  Dose 1: Unsolicited AEs: Mild | 3 | 6 | 94 | 88 | 6 | 4
  Dose 1: Unsolicited AEs: Moderate | 2 | 0 | 21 | 15 | 1 | 1
  Dose 1: Unsolicited AEs: Severe | 0 | 0 | 5 | 2 | 0 | 0
  Dose 2: Unsolicited AEs: number analyzed (Participants) | 4 | 3 | 77 | 75 | 10 | 7
  Dose 2: Unsolicited AEs: Mild | 4 | 1 | 54 | 63 | 9 | 1
  Dose 2: Unsolicited AEs: Moderate | 0 | 2 | 20 | 9 | 1 | 6
  Dose 2: Unsolicited AEs: Severe | 0 | 0 | 3 | 3 | 0 | 0

6. Primary Outcome: Number of Participants Who Experienced a Serious Adverse Event (SAE) During the Trial
Description: An SAE was defined as any untoward medical occurrence that, at any dose:
  * Resulted in death.
  * Was life-threatening.
  * Required inpatient hospitalization or prolongation of existing hospitalization.
  * Resulted in persistent disability/incapacity.
  * Was a congenital anomaly/birth defect in the offspring of the participant.
  * Was an important medical event.
  The Investigator assessed the relationship between trial vaccine and each occurrence of each AE.
Time Frame: Up to Day 393
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 6 μg: Aged 18-60 Years | CVnCoV 6 μg: Aged >60 Years | CVnCoV 12 μg: Aged 18-60 Years | CVnCoV 12 μg: Aged >60 Years | Active Control - Hepatitis A Vaccine: Aged 18-60 Years | Active Control - Pneumococcal Vaccine: Aged >60 Years
Number analyzed (Participants) | 12 | 11 | 289 | 295 | 31 | 30
Participants
  Any SAEs | 0 | 1 | 8 | 6 | 0 | 1
  Any related SAEs | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants Who Experienced an Adverse Event of Special Interest (AESI) During the Trial
Description: AESIs included:
  * AEs with a suspected immune-medicated etiology.
  * COVID-19 disease.
  * Other AEs relevant to SARS-CoV-2 vaccine development or the target disease.
  Participants who became unblinded and/or received a licensed/authorized vaccine were censored at the day after unblinding or at the day after receiving the licensed/authorized vaccine, whichever was earlier. The Investigator assessed the relationship between trial vaccine and each occurrence of each AE.
Time Frame: Up to Day 393
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 6 μg: Aged 18-60 Years | CVnCoV 6 μg: Aged >60 Years | CVnCoV 12 μg: Aged 18-60 Years | CVnCoV 12 μg: Aged >60 Years | Active Control - Hepatitis A Vaccine: Aged 18-60 Years | Active Control - Pneumococcal Vaccine: Aged >60 Years
Number analyzed (Participants) | 12 | 11 | 289 | 295 | 31 | 30
Participants
  Any AESIs | 1 | 3 | 36 | 23 | 7 | 3
  Any related AESIs | 0 | 0 | 0 | 1 | 0 | 0

8. Primary Outcome: Percentage of Participants Seroconverting for SARS-CoV-2 Spike Protein Receptor-Binding Domain (RBD) Antibodies on Day 29 and Day 43
Description: As measured by enzyme-linked immunosorbent assay (ELISA). In participants not exposed to SARS-CoV-2 before the trial seroconversion was defined as any increase in titer in antibodies against SARS-CoV-2 RBD versus baseline. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/authorized vaccine.
Time Frame: Baseline, Day 29 and Day 43
Population: The Immunogenicity Set including only participants who received Dose 1 and Dose 2 with no protocol deviations with impact to immunogenicity, who did not get exposed to SARS-CoV-2 before the trial, or during the trial before the applicable sample was collected and had a blood sample collected at Day 43.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CVnCoV 6 μg: Aged 18-60 Years | CVnCoV 6 μg: Aged >60 Years | CVnCoV 12 μg: Aged 18-60 Years | CVnCoV 12 μg: Aged >60 Years | Active Control - Hepatitis A Vaccine: Aged 18-60 Years | Active Control - Pneumococcal Vaccine: Aged >60 Years
Number analyzed (Participants) | 12 | 10 | 233 | 243 | 24 | 23
percentage of participants
  Day 29 | 0 [0.0 to 26.5] | 10.0 [0.3 to 44.5] | 11.6 [7.8 to 16.4] | 7.8 [4.8 to 11.9] | 0 [0.0 to 14.2] | 4.3 [0.1 to 21.9]
  Day 43: number analyzed (Participants) | 12 | 10 | 230 | 235 | 21 | 21
  Day 43 | 83.3 [51.6 to 97.9] | 80.0 [44.4 to 97.5] | 93.9 [90.0 to 96.6] | 80.9 [75.2 to 85.7] | 0 [0.0 to 16.1] | 4.8 [0.1 to 23.8]

9. Primary Outcome: Geometric Mean Titers (GMTs) of SARS-CoV-2 Spike Protein RBD Antibodies on Day 29 and Day 43
Description: As measured by ELISA. The SARS-CoV-2 spike RBD protein-specific antibodies are expressed as GMT (geometric mean of reciprocal duplicate dilutions). Concentration/titers marked as below the lower limit of quantification (LLOQ) were arbitrary replaced by half of the LLOQ for GMT computations purpose. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/authorized vaccine.
Time Frame: Day 29 and Day 43
Population: as for outcome 8
Measure: Geometric Mean (Standard Deviation); unit: titers
Arm/Group | CVnCoV 6 μg: Aged 18-60 Years | CVnCoV 6 μg: Aged >60 Years | CVnCoV 12 μg: Aged 18-60 Years | CVnCoV 12 μg: Aged >60 Years | Active Control - Hepatitis A Vaccine: Aged 18-60 Years | Active Control - Pneumococcal Vaccine: Aged >60 Years
Number analyzed (Participants) | 12 | 10 | 233 | 243 | 24 | 23
titers
  Day 29 | 50.000 (1.0000) | 57.154 (1.5264) | 67.221 (2.6624) | 63.828 (2.6005) | 56.724 (1.5434) | 52.112 (1.2195)
  Day 43: number analyzed (Participants) | 12 | 10 | 230 | 235 | 21 | 21
  Day 43 | 462.744 (3.4299) | 464.788 (4.2969) | 1733.125 (4.2886) | 552.782 (5.1208) | 57.455 (1.5663) | 62.667 (2.8146)

10. Primary Outcome: Percentage of Participants Seroconverting for SARS-CoV-2 Neutralizing Antibodies on Day 29 and Day 43
Description: As measured by an activity assay. In participants not exposed to SARS-CoV-2 before the trial, seroconversion was defined as any increase in titer in SARS-CoV-2 neutralizing antibodies versus baseline. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/ authorized vaccine.
Time Frame: Baseline, Day 29 and Day 43
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CVnCoV 6 μg: Aged 18-60 Years | CVnCoV 6 μg: Aged >60 Years | CVnCoV 12 μg: Aged 18-60 Years | CVnCoV 12 μg: Aged >60 Years | Active Control - Hepatitis A Vaccine: Aged 18-60 Years | Active Control - Pneumococcal Vaccine: Aged >60 Years
Number analyzed (Participants) | 12 | 10 | 180 | 154 | 15 | 16
percentage of participants
  Day 29 | 0 [0.0 to 26.5] | 0 [0.0 to 30.8] | 8.3 [4.7 to 13.4] | 7.8 [4.1 to 13.2] | 0 [0.0 to 21.8] | 0 [0.0 to 20.6]
  Day 43: number analyzed (Participants) | 12 | 10 | 177 | 153 | 13 | 15
  Day 43 | 66.7 [34.9 to 90.1] | 70.0 [34.8 to 93.3] | 86.4 [80.5 to 91.1] | 77.1 [69.6 to 83.5] | 0 [0.0 to 24.7] | 0 [0.0 to 21.8]

11. Primary Outcome: GMTs of SARS-CoV-2 Neutralizing Antibodies on Day 29 and Day 43
Description: The SARS-CoV-2 neutralizing antibodies are expressed as GMT (geometric mean of reciprocal duplicate dilutions). Concentration/titers marked as below the lower limit of quantification (LLOQ) were arbitrary replaced by half of the LLOQ for GMT computations purpose. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/authorized vaccine.
Time Frame: Day 29 and Day 43
Population: as for outcome 8
Measure: Geometric Mean (Standard Deviation); unit: titers
Arm/Group | CVnCoV 6 μg: Aged 18-60 Years | CVnCoV 6 μg: Aged >60 Years | CVnCoV 12 μg: Aged 18-60 Years | CVnCoV 12 μg: Aged >60 Years | Active Control - Hepatitis A Vaccine: Aged 18-60 Years | Active Control - Pneumococcal Vaccine: Aged >60 Years
Number analyzed (Participants) | 12 | 10 | 180 | 154 | 15 | 16
titers
  Day 29 | 5.000 (1.0000) | 5.000 (1.0000) | 5.912 (2.0106) | 6.234 (2.4723) | 5.000 (1.0000) | 5.000 (1.0000)
  Day 43: number analyzed (Participants) | 12 | 10 | 177 | 153 | 13 | 15
  Day 43 | 16.339 (3.6716) | 20.705 (2.8993) | 50.298 (4.0175) | 26.848 (3.9517) | 5.000 (1.0000) | 5.000 (1.0000)

12. Secondary Outcome: Number of Participants Who Experienced a Solicited Adverse Event (AE) Occurring on the Day of Booster Vaccination and the Following 7 Days
Description: as for outcome 1
Time Frame: Up to 7 days after booster vaccination (Days 57 to 64 and Days 180 to 187)
Population: Safety Analysis Set: All participants who received at least 1 dose of trial vaccine and for whom any post-vaccination safety data are available. Only participants who received a booster vaccination on Day 57 or Day 180 and had evaluable samples at each visit were included.
Measure: Count of Participants; unit: Participants
Groups:
- CVnCoV 12 μg: Aged >60 Years - Day 57 Booster: Participants in Part 1 and Part 2 were administered a booster vaccination with CVnCoV 12 μg as an intramuscular injection by needle in the deltoid area on Day 57. Participants in this group were aged over 60 years old.
- CVnCoV 12 μg: Aged 18-60 Years - Day 180 Booster: Participants in Part 1 and Part 2 were administered a booster vaccination with CVnCoV 12 μg as an intramuscular injection by needle in the deltoid area on Day 180. Participants in this group were between the ages of 18 to 60 years old.
- CVnCoV 12 μg: Aged >60 Years - Day 180 Booster: Participants in Part 1 and Part 2 were administered a booster vaccination with CVnCoV 12 μg as an intramuscular injection by needle in the deltoid area on Day 180. Participants in this group were aged over 60 years old.
Arm/Group | CVnCoV 12 μg: Aged >60 Years - Day 57 Booster | CVnCoV 12 μg: Aged 18-60 Years - Day 180 Booster | CVnCoV 12 μg: Aged >60 Years - Day 180 Booster
Number analyzed (Participants) | 30 | 30 | 15
Participants
  Any solicited local AEs | 15 | 24 | 12
  Any solicited systemic AEs | 15 | 24 | 8
  Any related solicited systemic AEs | 15 | 24 | 8

13. Secondary Outcome: Intensity of Solicited AEs Per FDA Toxicity Grading Scale Occurring on the Day of Booster Vaccination and the Following 7 Days
Description: as for outcome 2
Time Frame: Up to 7 days after booster vaccination (Days 57 to 64 and Days 180 to 187)
Population: The Safety Analysis Set including only participants who experienced solicited local and systemic AEs. Only participants who received a booster vaccination on Day 57 or Day 180 and had evaluable samples at each visit were included.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg: Aged >60 Years - Day 57 Booster | CVnCoV 12 μg: Aged 18-60 Years - Day 180 Booster | CVnCoV 12 μg: Aged >60 Years - Day 180 Booster
Number analyzed (Participants) | 15 | 24 | 12
Participants
  Any solicited local AEs: Grade 1 | 14 | 18 | 9
  Any solicited local AEs: Grade 2 | 1 | 5 | 3
  Any solicited local AEs: Grade 3 | 0 | 1 | 0
  Any solicited systemic AEs: number analyzed (Participants) | 15 | 24 | 8
  Any solicited systemic AEs: Grade 1 | 13 | 11 | 6
  Any solicited systemic AEs: Grade 2 | 2 | 12 | 2
  Any solicited systemic AEs: Grade 3 | 0 | 1 | 0

14. Secondary Outcome: Duration of Solicited AEs Occurring on the Day of Booster Vaccination and the Following 7 Days
Description: Solicited local AEs (injection site pain, redness, swelling, and itching) and solicited systemic AEs (fever, headache, fatigue, chills, myalgia, arthralgia, nausea/vomiting, and diarrhea) were recorded on the day of vaccination and the following 7 days using a diary (electronic or paper). Duration is calculated as consecutive days with a respective solicited AE regardless of the grade of the adverse event.
Time Frame: Up to 7 days after booster vaccination (Days 57 to 64 and Days 180 to 187)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CVnCoV 12 μg: Aged >60 Years - Day 57 Booster | CVnCoV 12 μg: Aged 18-60 Years - Day 180 Booster | CVnCoV 12 μg: Aged >60 Years - Day 180 Booster
Number analyzed (Participants) | 15 | 24 | 12
days
  Any solicited local AEs | 1.7 (0.80) | 2.0 (1.53) | 1.6 (0.79)
  Any solicited systemic AEs: number analyzed (Participants) | 15 | 24 | 8
  Any solicited systemic AEs | 2.8 (2.18) | 2.0 (1.71) | 2.0 (2.07)

15. Secondary Outcome: Number of Participants Who Experienced an Unsolicited AE Occurring on the Day of Booster Vaccination and the Following 28 Days
Description: as for outcome 4
Time Frame: Up to 28 days after booster vaccination (Days 57 to 85 and Days 180 to 208)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg: Aged >60 Years - Day 57 Booster | CVnCoV 12 μg: Aged 18-60 Years - Day 180 Booster | CVnCoV 12 μg: Aged >60 Years - Day 180 Booster
Number analyzed (Participants) | 30 | 30 | 15
Participants
  Any unsolicited AEs | 7 | 6 | 2
  Any related unsolicited AEs | 1 | 4 | 2

16. Secondary Outcome: Intensity of Unsolicited AEs Per the Investigator's Assessment Occurring on the Day of Booster Vaccination and the Following 28 Days
Description: as for outcome 5
Time Frame: Up to 28 days after booster vaccination (Days 57 to 85 and Days 180 to 208)
Population: The Safety Analysis Set including only participants who experienced unsolicited AEs. Only participants who received a booster vaccination on Day 57 or Day 180 and had evaluable samples at each visit were included.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg: Aged >60 Years - Day 57 Booster | CVnCoV 12 μg: Aged 18-60 Years - Day 180 Booster | CVnCoV 12 μg: Aged >60 Years - Day 180 Booster
Number analyzed (Participants) | 7 | 6 | 2
Participants
  Mild | 6 | 5 | 2
  Moderate | 1 | 0 | 0
  Severe | 0 | 1 | 0

17. Secondary Outcome: Percentage of Participants Seroconverting for SARS-CoV-2 Spike Protein RBD Antibodies on Day 57, Day 85, Day 180, Day 208 and Day 393
Description: As measured by ELISA. In participants not exposed to SARS-CoV-2 before the trial seroconversion was defined as any increase in titer in antibodies against SARS-CoV-2 RBD versus baseline. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/ authorized vaccine.
Time Frame: For participants who received the booster vaccination on Day 57: Baseline, Day 57, Day 85 and Day 180. For participants who received the booster vaccination on Day 180: Baseline, Day 180, Day 208 and Day 393
Population: The Immunogenicity Set including only participants who received Dose 1, Dose 2 and a booster dose on Day 57 or Day 180 with no protocol deviations with impact to immunogenicity, who did not get exposed to SARS-CoV-2 before the trial, or during the trial before the applicable sample was collected and had a blood sample collected at Day 43.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- CVnCoV 12 μg: Aged >60 Years - Day 57 Booster: Participants in Part 1 were administered a booster vaccination with CVnCoV 12 μg as an intramuscular injection by needle in the deltoid area on Day 57. Participants in this group were aged over 60 years old.
- CVnCoV 12 μg: Aged 18-60 Years - Day 180 Booster: Participants in Part 1 were administered a booster vaccination with CVnCoV 12 μg as an intramuscular injection by needle in the deltoid area on Day 180. Participants in this group were between the ages of 18 to 60 years old.
- CVnCoV 12 μg: Aged >60 Years - Day 180 Booster: Participants in Part 1 were administered a booster vaccination with CVnCoV 12 μg as an intramuscular injection by needle in the deltoid area on Day 180. Participants in this group were aged over 60 years old.
Arm/Group | CVnCoV 12 μg: Aged >60 Years - Day 57 Booster | CVnCoV 12 μg: Aged 18-60 Years - Day 180 Booster | CVnCoV 12 μg: Aged >60 Years - Day 180 Booster
Number analyzed (Participants) | 28 | 21 | 13
percentage of participants
  Day 57: number analyzed (Participants) | 28 | 0 | 0
  Day 57 | 82.1 [63.1 to 93.9] |  |
  Day 85: number analyzed (Participants) | 25 | 0 | 0
  Day 85 | 100 [86.3 to 100] |  |
  Day 180: number analyzed (Participants) | 21 | 21 | 13
  Day 180 | 100 [83.9 to 100] | 90.5 [69.6 to 98.8] | 69.2 [38.6 to 90.9]
  Day 208: number analyzed (Participants) | 0 | 20 | 10
  Day 208 |  | 100 [83.2 to 100] | 100 [69.2 to 100]
  Day 393: number analyzed (Participants) | 0 | 1 | 0
  Day 393 |  | 100 [2.5 to 100] |

18. Secondary Outcome: GMTs of SARS-CoV-2 Spike Protein RBD Antibodies on Day 57, Day 85, Day 180, Day 208 and Day 393
Description: As measured by ELISA. The SARS-CoV-2 spike RBD protein-specific antibodies are expressed as GMT (geometric mean of reciprocal duplicate dilutions). Concentration/titers marked as below the lower limit of quantification (LLOQ) were arbitrary replaced by half of the LLOQ for GMT computations purpose. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/ authorized vaccine.
Time Frame: For participants who received the booster vaccination on Day 57: Day 57, Day 85 and Day 180. For participants who received the booster vaccination on Day 180: Day 180, Day 208 and Day 393
Population: as for outcome 17
Measure: Geometric Mean (Standard Deviation); unit: titers
Arm/Group | CVnCoV 12 μg: Aged >60 Years - Day 57 Booster | CVnCoV 12 μg: Aged 18-60 Years - Day 180 Booster | CVnCoV 12 μg: Aged >60 Years - Day 180 Booster
Number analyzed (Participants) | 28 | 21 | 13
titers
  Day 57: number analyzed (Participants) | 28 | 0 | 0
  Day 57 | 516.198 (4.6157) |  |
  Day 85: number analyzed (Participants) | 25 | 0 | 0
  Day 85 | 2889.963 (2.9473) |  |
  Day 180: number analyzed (Participants) | 21 | 21 | 13
  Day 180 | 1449.055 (2.1869) | 445.661 (3.1744) | 153.160 (2.8146)
  Day 208: number analyzed (Participants) | 0 | 20 | 10
  Day 208 |  | 10094.652 (2.1020) | 4153.249 (2.2450)
  Day 393: number analyzed (Participants) | 0 | 1 | 0
  Day 393 |  | 915.460 (NA) — Standard deviation was not estimable as only 1 participant had available data. |

19. Secondary Outcome: Percentage of Participants Seroconverting for SARS-CoV-2 Neutralizing Antibodies on Day 57, Day 85, Day 180, Day 208 and Day 393
Description: As measured by an activity assay. In participants not exposed to SARS-CoV-2 before the trial, seroconversion was defined as any increase in titer in SARS-CoV-2 neutralizing antibodies versus baseline. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/authorized vaccine.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CVnCoV 12 μg: Aged >60 Years - Day 57 Booster | CVnCoV 12 μg: Aged 18-60 Years - Day 180 Booster | CVnCoV 12 μg: Aged >60 Years - Day 180 Booster
Number analyzed (Participants) | 28 | 21 | 13
percentage of participants
  Day 57: number analyzed (Participants) | 28 | 0 | 0
  Day 57 | 75.0 [55.1 to 89.3] |  |
  Day 85: number analyzed (Participants) | 25 | 0 | 0
  Day 85 | 96.0 [79.6 to 99.9] |  |
  Day 180: number analyzed (Participants) | 21 | 21 | 13
  Day 180 | 57.1 [34.0 to 78.2] | 28.6 [11.3 to 52.2] | 7.7 [0.2 to 36.0]
  Day 208: number analyzed (Participants) | 0 | 20 | 10
  Day 208 |  | 100 [83.2 to 100] | 90.0 [55.5 to 99.7]
  Day 393: number analyzed (Participants) | 0 | 1 | 0
  Day 393 |  | 100 [2.5 to 100] |

20. Secondary Outcome: GMTs of SARS-CoV-2 Neutralizing Antibodies on Day 57, Day 85, Day 180, Day 208 and Day 393
Description: As measured by an activity assay. The SARS-CoV-2 neutralizing antibodies are expressed as GMT (geometric mean of reciprocal duplicate dilutions). Concentration/titers marked as below the lower limit of quantification (LLOQ) were arbitrary replaced by half of the LLOQ for GMT computations purpose. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/ authorized vaccine.
Time Frame: as for outcome 18
Population: as for outcome 17
Measure: Geometric Mean (Standard Deviation); unit: titers
Arm/Group | CVnCoV 12 μg: Aged >60 Years - Day 57 Booster | CVnCoV 12 μg: Aged 18-60 Years - Day 180 Booster | CVnCoV 12 μg: Aged >60 Years - Day 180 Booster
Number analyzed (Participants) | 28 | 21 | 13
titers
  Day 57: number analyzed (Participants) | 28 | 0 | 0
  Day 57 | 25.937 (4.4384) |  |
  Day 85: number analyzed (Participants) | 25 | 0 | 0
  Day 85 | 74.642 (3.0879) |  |
  Day 180: number analyzed (Participants) | 21 | 21 | 13
  Day 180 | 16.957 (3.3656) | 7.308 (2.5328) | 5.867 (1.7802)
  Day 208: number analyzed (Participants) | 0 | 20 | 10
  Day 208 |  | 141.724 (2.0232) | 54.639 (3.3018)
  Day 393: number analyzed (Participants) | 0 | 1 | 0
  Day 393 |  | 28.280 (NA) — Standard deviation was not estimable as only 1 participant had available data. |

ADVERSE EVENTS:
Time Frame: Day 1 to Day 393
Description: Adverse events were collected based on intervention type and were not collected separately for the active control arm.
Groups:
- CVnCoV 6 μg: Participants in Part 1 were vaccinated with CVnCoV 6 μg as an intramuscular injection by needle in the deltoid area on Day 1 and Day 29.
- CVnCoV 12 μg: Participants in Part 1 and Part 2 were vaccinated with CVnCoV 12 μg as an intramuscular injection by needle in the deltoid area on Day 1 and Day 29.
  CVnCoV was administered again as a booster vaccination on Day 57 or Day 180 in a sub-group of participants in Part 1.
- Active Control: Participants in Part 1 and Part 2 were vaccinated with an active control (hepatitis A vaccine if aged 18-60 years old or pneumococcal vaccine if aged over 60 years old) as an intramuscular injection by needle in the deltoid area on Day 1 and Day 29.
Arm/Group | CVnCoV 6 μg | CVnCoV 12 μg | Active Control
All-Cause Mortality (participants affected / at risk) | 0/23 | 3/584 | 1/61
Serious Adverse Events (participants affected / at risk) | 1/23 | 14/584 | 1/61
Other Adverse Events (participants affected / at risk) | 21/23 | 567/584 | 59/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CVnCoV 6 μg (N=23) | CVnCoV 12 μg (N=584) | Active Control (N=61)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CVnCoV 6 μg (N=23) | CVnCoV 12 μg (N=584) | Active Control (N=61)
Injection site pain (General disorders) | 17 (30) | 526 (1012) | 47 (75)
Fatigue (General disorders) | 7 (16) | 315 (555) | 22 (29)
Chills (General disorders) | 8 (13) | 254 (384) | 10 (12)
Pyrexia (General disorders) | 4 (4) | 182 (233) | 4 (6)
Swelling (General disorders) | 2 (2) | 52 (60) | 8 (8)
Discomfort (General disorders) | 3 (3) | 15 (18) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 10 (10) | 4 (4)
Headache (Nervous system disorders) | 13 (24) | 390 (763) | 33 (46)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 315 (505) | 13 (21)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (15) | 237 (362) | 12 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 46 (54) | 3 (3)
Nasopharyngitis (Infections and infestations) | 4 (5) | 155 (217) | 12 (14)
COVID-19 (Infections and infestations) | 3 (3) | 108 (109) | 12 (12)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 68 (79) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (3) | 14 (14) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 107 (140) | 6 (6)
Nausea (Gastrointestinal disorders) | 2 (2) | 69 (83) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 45 (58) | 5 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 52 (66) | 11 (12)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 31 (34) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 31 (31) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 16 (17) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 14 (14) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 15 (15) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/47/NCT04515147/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT04515147/SAP_001.pdf